CLINICAL TRIAL: NCT02081313
Title: Syndrome de Netherton : Aspects Cliniques, Physiopathologiques et Identification de Cibles thérapeutiques
Brief Title: Natural History and Biological Study of Netherton Syndrome
Acronym: NSnatbio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: C12-56; 2013-A00275-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Netherton Syndrome; Healthy
Keywords: Netherton syndrome; Immune system; Skin barrier
MeSH Terms: conditions — Netherton Syndrome | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Netherton syndrome (Active Comparator): Patients with Netherton syndrome
  Interventions: Other: Biopsy; Other: Blood sample
- Healthy controls (Active Comparator): healthy controls
  Interventions: Other: Biopsy; Other: Blood sample

INTERVENTIONS:
Other: Biopsy
Other: Blood sample

SUMMARY:
This study aims at studying the natural history of Netherton syndrome (NS), to identify the consequences of LEKTI deficiency on the immune system and to characterize new molecular mechanisms involved in the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child (no age limit)
* Confirmed diagnosis of Netherton syndrome
* Signed informed consent form for the patient or his legal representative

Exclusion Criteria:

* Bleeding disorder precluding skin biopsy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09-04 (Actual)

PRIMARY OUTCOMES:
Measurement of seric cytokines levels | 3 months after patient recruitment

SECONDARY OUTCOMES:
Pattern of skin abnormalities | 3 months after patient recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hovnanian, MD, PhD, Principal Investigator — INSERM U1163
Locations (1):
- Imagine Institute for genetic diseases, Paris, France

REFERENCES:
- [Result] Barbieux C, Bonnet des Claustres M, Fahrner M, Petrova E, Tsoi LC, Gouin O, Leturcq F, Nicaise-Roland P, Bole C, Beziat V, Bourrat E, Schilling O, Gudjonsson JE, Hovnanian A. Netherton syndrome subtypes share IL-17/IL-36 signature with distinct IFN-alpha and allergic responses. J Allergy Clin Immunol. 2022 Apr;149(4):1358-1372. doi: 10.1016/j.jaci.2021.08.024. Epub 2021 Sep 17. PMID 34543653
- [Result] Petrova E, Duthoit A, Prassas I, Hovnanian A. Unveiling serine protease activity profiles in Netherton syndrome skin across clinical subtypes by noninvasive analysis. Am J Physiol Cell Physiol. 2025 Oct 1;329(4):C1139-C1149. doi: 10.1152/ajpcell.01027.2024. Epub 2025 Sep 4. PMID 40908106